CLINICAL TRIAL: NCT03210727
Title: A Mixed Methods Descriptive Study Exploring the Needs and Preferences of Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: CAREgiver Study for Patients Undergoing HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D17033
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a single arm design will be used to pilot test the Ready to CARE program with 20 caregivers (while also measuring outcomes in the 20 patients receiving HSCT)..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): This arm will be used to pilot test the Ready to CARE program (with the caregivers) and measure outcomes (in the patients).
  Interventions: Behavioral: Ready to CARE program

INTERVENTIONS:
Behavioral: Ready to CARE program — The intervention is built upon a model of caregiver well-being that identifies four domains of quality of life: physical, psychological, social, and spiritual well-being. For each domain, there are stressors (i.e., factors that make it hard to be a caregiver) and buffers (i.e., factors that help people be effective caregivers). Our Ready to CARE intervention begins by presenting caregivers with the model in order to generate a profile of personal stressors and buffers. From there, caregivers select from a "menu" of strategies that can be used to minimize stressors and create buffers in their daily life. The investigators will have six 45-minute sessions with the caregivers that will primarily occur while the patient is admitted for stem cell reinfusion.

SUMMARY:
The investigators will use a single arm design and deliver a new supportive intervention entitled, "Ready to Connect, Actively Relax and Exercise (CARE)." The purpose of the study is to describe the feasibility, acceptability, and potential effectiveness of the Ready to CARE intervention. Effectiveness outcomes include caregiver self-efficacy, distress, and coping style, and patient quality of life, symptom burden, and healthcare utilization.

DETAILED DESCRIPTION:
During the first phase of this study, the investigators enrolled caregivers of patients undergoing hematopoietic stem cell transplantation (HSCT) into a descriptive study. The investigators used quantitative and qualitative measures to describe the caregivers self-efficacy, distress, and coping style, and solicit their opinions about how to improve our supportive care for caregivers.

Informed by those data, the investigators now will study the effectiveness of the supportive intervention.

The long-term goal of this research is to develop a pragmatic, replicable intervention that supports caregivers and promotes the health and well-being of the caregiver-HSCT patient dyad.

ELIGIBILITY:
Inclusion Criteria:

* Providing informal, unpaid care for a person who is 18 years of age or older and is scheduled to receive an allogeneic or autologous HSCT within the next three months.
* The caregiver's loved one ("patient") undergoing the transplant will be asked to enroll in the study to provide data regarding quality of life and symptom burden and to allow access of the medical record to ascertain healthcare utilization data. (Caregivers will not be excluded from the study if the patient declines to enroll.)

Exclusion Criteria:

* Under the age of 18 for either caregiver or patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Enrollment statistics | Throughout the study, an average of one year
  Number enrolled in study divided by number eligible

SECONDARY OUTCOMES:
Retention | Throughout the study, an average of one year
  number completing all study assessments divided by number enrolled
Goal Attainment | Day 30 after stem cell reinfusion
  average goal attainment score between sessions
Session Completion | Day 30 after stem cell reinfusion
  Average number of sessions completed
Caregiver Satisfaction | Day 30 after stem cell reinfusion
  Average score on satisfaction survey
Caregiver Self-efficacy | Day 100 after stem cell reinfusion
  Average change score on Caregiver Self-efficacy Scale
Caregiver Coping style | Day 100 after stem cell reinfusion
  Average change score on Brief Cope
Patient Quality of Life | Day 100 after stem cell reinfusion
  Average change score on Functional Assessment of Cancer Therapy- Bone Marrow Transplant
Patient symptom burden | Day 100 after stem cell reinfusion
  Average change score on MD Anderson Symptom Inventory
Patient healthcare utilization | Day 100 after stem cell reinfusion
  Average number of re-hospitalizations, urgent care or emergency department visits, and telephone calls to bone marrow transplant program

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen D Lyons, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No